CLINICAL TRIAL: NCT01145963
Title: Understanding Pasta Formulations on Satiation in Healthy Weight Women
Brief Title: Pasta Formulations and Their Effect on Appetite
Acronym: SAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Collaborators: Barilla America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: SAT 2010-042
Record Dates: First submitted 2010-06-15; First posted 2010-06-17 (Estimated); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Appetite
Keywords: pasta; appetite; hunger; satiation; nutrition; Psychological Phenomena and Processes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- experimental pasta B (Experimental): Past B
  Interventions: Other: Experimental pasta B
- experimental pasta C (Experimental): Pasta C
  Interventions: Other: Experimental pasta C
- Control pasta (Placebo Comparator): Control
  Interventions: Other: Control pasta

INTERVENTIONS:
Other: Control pasta — control pasta
  Arms: Control pasta
Other: Experimental pasta B — experimental pasta
  Arms: experimental pasta B
Other: Experimental pasta C — experimental pasta
  Arms: experimental pasta C

SUMMARY:
Investigators are interested in learning how appetite responds to pasta containing different amounts of protein and fiber. In this research study, subjects will be asked to eat as much as they want of pasta containing different amounts of protein and fiber mixtures, thereafter subjects will describe their feelings of hunger, fullness and desire to eat for 3 hours afterwards. Subjects will be asked to do this on three separate occasions.

DETAILED DESCRIPTION:
The study is a randomized, 3-arm, treatment-controlled, within-subjects, 3-hour postprandial crossover study to evaluate the satiation effects of pasta formulations on lunch intake in healthy weight women. The study design will test 3 varying pasta formulations (2 experimental and 1 standard control) in a lunch setting in relatively healthy unrestrained women.

This study will require one initial screening visit (approximately 1 hour) and three study visits each lasting approximately 4 hours. All visits should be done in 1 month. We are looking for healthy, non-smoking women older than 18 years of age with no significant medical history.

The initial screening visit will determine subject eligibility through height, weight and waist circumference measurements, blood glucose test (finger prick) and eating, health, exercise and mood surveys.

If willing and eligible to participate, subjects will have 3 study visits. At each visits, subjects will be asked to consume as much as they would like of the pasta meal and beverage in a lunch setting and thereafter will be followed for 3 hours assessing subjective feelings of satiety. The lunch meal will be provided 5 hours after a standardized breakfast (usual breakfast for each subject at the same time of day on each study visit day). During the course of the study, subjects will be instructed to maintain their usual level of activity and diet. Four day food records will be maintained throughout the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Females
* 18 years of age and older
* Body mass index (BMI) between 18.5 and 24.9 kg/m2, inclusive
* No clinical evidence of cardiovascular, metabolic, respiratory, renal, gastrointestinal or hepatic disease
* Unrestrained eater (score < 10 on the Three Factor Eating Questionnaire)

Exclusion Criteria:

* Pregnant and/or lactating or planning for pregnancy
* Allergies or intolerances to foods consumed in the study
* Fasting blood glucose > 110 mg/dL. Subjects identified with elevated fasting blood glucose levels will be will be advised to contact their primary care physician for appropriate follow-up care.
* Taking over the counter fiber supplements or other supplements that may interfere with the study procedures or endpoints
* Taking prescription medications that may interfere with study procedures or endpoints ( medications that affect appetite)
* Subjects with unusual dietary habits (e.g. pica)
* Actively losing weight or trying to lose weight (unstable body weight fluctuations of > 5 kg in a 60 day period)
* Excessive exercisers or trained athletes
* Addicted to drugs and/or alcohol
* Medically documented psychiatric or neurological disturbances
* Smoker (past smoker may be allowed if cessation is > 2 years)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-06-01 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

PRIMARY OUTCOMES:
To investigate the effect of pasta formulations incorporated into a lunch meal on satiation (meal termination) as determined by energy intake of the meal along with subjective responses on visual analog scales and subsequent food intake. | 3 hour post prandial study
  Meals will be provided 4 1/2 hours after a standardized breakfast (subject's own usual breakfast in the same quantity at the same time before each study visit) and subjects will be able to eat as much of the pasta as they would like and may request more if desired. Immediately thereafter, subjects will record satiety responses at 0 min (immediately post consumption), 20, 40, 60, 90, 120, 150 and 180 on a visual analog scale (VAS). The subject will answer a series of questions on the VAS at each respective time point describing their feelings of hunger, fullness and desire to eat.

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, PhD, MS, Principal Investigator — Clinical Nutrition Research Center, Illinois Institute of Technology; Indika Edirisinghe, PhD, Principal Investigator — Clinical Nutrition Research Center, Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States